CLINICAL TRIAL: NCT04097704
Title: An Observational Follow-on Study to Describe the Pharmacogenetics of the CC-90007-CP-003 Study Cohort
Brief Title: Pharmacogenetics Sampling of the CC-90007-CP-003 Study Cohort
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NDS-CP-003; U1111-1237-0411 (Other: WHO)
Record Dates: First submitted 2019-09-19; First posted 2019-09-20 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Hepatic Insufficiency
Keywords: Hepatic impairment; CC-90007-CP-003; Healthy Subject
MeSH Terms: conditions — Hepatic Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a multi-center observational follow-up study to collect saliva samples that allow pharmacogenetic analysis of the subjects that participated in the CC-90007-CP-003 study.

Approximately 28 subjects with moderate and severe hepatic impairment and healthy control subjects with normal hepatic function will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

Each subject must satisfy all of the following criteria to be enrolled in this study:

1. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
2. Subject is able to communicate with the Investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules and other protocol requirements.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Subject participated in the CC-90007-CP-003 study.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any condition which places the subject at unacceptable risk if he/she were to participate in the study.
2. Subject has any condition that confounds the ability to interpret data from the study.

Sponsor's medical monitor should be consulted on suspected conditions under this exclusion criterion, prior to exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 28 subjects from the CC-90007-CP-003 study (from any race, males or non-pregnant and non-nursing females) will be enrolled. The study will be conducted at approximately 3 sites in the US that participated in the CC-90007-CP-003 study. Subjects may not be replaced with subjects that did not participate in the CC-90007-CP-003 study.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects whose primary saliva sample yields DNA that meets modified PharmacoScan® workflow acceptability criteria | Day 1
  DNA Quality

SECONDARY OUTCOMES:
Adverse Events (AEs) | Time from ICF to Day 1
  Number of participants with adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Leon Carayannopoulos, MD, Study Director — Celgene Corporation
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Orlando Clinical Research Center OCRC, Orlando, Florida
  - Volunteer Research Group and New Orleans Center for Clinical Research - Knoxville, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/